CLINICAL TRIAL: NCT05637580
Title: Real-world Analysis of Pathological Tumor and Lymph Node Responses After Neoadjuvant Immunochemotherapy in Initially-unresectable Non-small Cell Lung Cancer
Brief Title: Pathological Tumor and Lymph Node Responses After Neoadjuvant Immunochemotherapy in Initially-unresectable NSCLC
Status: Completed | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LUNGTN
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Non Small Cell Lung Cancer; Immunotherapy; Chemotherapy; Tumour, Residual
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- combined well responder: Both primary tumor and nodal response achieve major pathological response (MPR).
  Interventions: Drug: Timing of drug administration
- poor responder: Primary tumor or/and nodal response can not achieve MPR.
  Interventions: Drug: Timing of drug administration

INTERVENTIONS:
Drug: Timing of drug administration — The effect of drug administration timing on tumor and lymph node responses was observed.

SUMMARY:
This is a real-world study with the largest sample size investigating the pathological tumor and lymph node responses to neoadjuvant immunochemotherapy in non-small cell lung cancer to date. Patients with initially unresectable NSCLC underwent immunochemotherapy and response to treatment was assessed after every two treatment cycles. Clinicopathologic features of patients including epidemiological data, clinical manifestations, operation strategies, pathological findings, and prognostic information were recorded and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage III NSCLC who received neoadjuvant immunochemotherapy.
* early-stage NSCLC patients who were initially unresectable.
* 18 years of age or older.
* Karnofsky performance status (KPS) score of 100 or 90.

Exclusion Criteria:

* Patients with stage IV NSCLC
* Patients with known ALK translocations or EGFR mutations.
* Karnofsky performance status (KPS) score <90.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage II-III NSCLC who received neoadjuvant immunochemotherapy (time) in Guangdong Provincial People's Hospital were eligible for this study. We also included early-stage NSCLC patients who were unsuitable or unable to tolerate surgery after first evaluation. Eligible patients were 18 years of age or older, had a karnofsky performance status (KPS) score of 100 or 90 (on a scale from 0 to 100 with higher score indicating better ability to carry out daily activities). Patients with distant tumor metastasis or with known ALK translocations or EGFR mutations were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Event-free survival | At least one year
  the time from diagnosis to any progression of disease precluding surgery, progression or recurrence of disease after surgery or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Guibin Qiao, MD, Study Director — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China